CLINICAL TRIAL: NCT06142916
Title: THE EFFECT OF TRAINING PROVIDED WITH VIRTUAL REALITY ON NURSES' MENTAL HEALTH LITERACY AND STIGMA LEVEL TOWARDS MENTAL DISEASES
Brief Title: The Effect of Virtual Reality Training on Mental Health Literacy and Stigma
Acronym: MHLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Melek Sahan, postrgraduate student, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2032
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Disorder; Literacy; Stigma, Social
Keywords: Mental Health Disorder; Mental Health Literacy; Stigma; Virtual Reality
MeSH Terms: conditions — Mental Disorders; Literacy; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHLS (Experimental)
  Interventions: Other: Vırtual Realıty Traınıng On Mental Health Lıteracy And Stıgma
- CONTROL GROUP (Active Comparator)
  Interventions: Other: Classical Education

INTERVENTIONS:
Other: Vırtual Realıty Traınıng On Mental Health Lıteracy And Stıgma — Nurses in the intervention group will be taken to a suitable room on the ward and virtual reality glasses will be worn. Mental health literacy training prepared by researchers by scanning the literature will be given using virtual reality glasses. Educational content; definition of mental health, definition of mental illness, definition and importance of mental health literacy, the most common mental illnesses in hospitals, Schizophrenia, Depression, Bipolar Disorder, Anxiety Disorders, Obsessive Compulsive Disorder (OCD), Post-Traumatic Stress Disorder (PTSD), Substance Use Disorder , Suicide-Self-Harm, Mental Health Literacy and Stigma, and where to find resources to obtain information about mental health. Information about the diagnostic criteria, risk factors, treatment methods, and what to pay attention to for the diseases discussed will be given. Animations will be prepared for each topic. The training is planned to last 45 minutes.
  Arms: MHLS
Other: Classical Education — Nurses in the control group will be given mental health literacy training using the classical method using brochures. Educational content; definition of mental health, definition of mental illness, definition and importance of mental health literacy, the most common mental illnesses in hospitals, Schizophrenia, Depression, Bipolar Disorder, Anxiety Disorders, Obsessive Compulsive Disorder (OCD), Post-Traumatic Stress Disorder (PTSD), Substance Use Disorder , Suicide-Self-Harm, Mental Health Literacy and Stigma, and where to find resources to obtain information about mental health. Information about the diagnostic criteria, risk factors, treatment methods, and what to pay attention to for the diseases discussed will be given. The training is planned to last 45 minutes.
  Arms: CONTROL GROUP

SUMMARY:
Purpose: This study will be conducted to examine the effect of virtual reality training on nurses' mental health literacy and stigma level towards mental illnesses.

Design: The study is a randomized controlled experimental research. Method: The population of the research consists of 110 nurses working in a public hospital. Power analysis was performed with G* Power software to determine the number of nurses constituting the research sample. The sample size was determined as 25 people in each group. Considering that there may be data loss in the study, it is planned to include 30 people in the intervention group and 30 people in the control group. Nurses who volunteer to participate in the study and fill out the pre-test will be randomly assigned to the groups using the Statistical Analysis Software program to ensure random distribution to the intervention and control groups. Personal Information Form, Mental Health Literacy Scale (MHLS) and Opening Minds Stigma Scale for Healthcare Providers (OMS-HC) will be used in study data collection.

Hypotheses:

H1: The mental health literacy level of nurses who receive training with virtual reality is higher than nurses who receive classical training.

H2: The level of stigmatization towards mental illnesses of nurses trained with virtual reality is lower than nurses who received classical training.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Becoming a nurse
* Being actively working in a public hospital in Istanbul
* Volunteering to participate in the study
* Not having worked in a psychiatric ward before

Exclusion Criteria:

Being under 18 years of age

* Not being a nurse
* Not actively working in the hospital where the study will be conducted
* Not volunteering to participate in the study
* Having worked in a psychiatric ward before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | For 2 weeks
  n the form prepared by the researchers in line with the literature, the nurses' introductory information; age, gender, marital status, education level, income level, unit of employment, working period, status of receiving psychiatric help, status of having a family member with a mental disorder, status of obtaining information about mental health, sources from which they obtained information about mental health and mental health. There are a total of 11 questions, including the status of receiving literacy education.
Mental Health Literacy Scale | For 2 weeks
  The scale, which was developed by O'Connor and Casey (2015) and whose Turkish validity and reliability study was conducted by Kesgin et al. (2020), consists of 35 items. The maximum score is 160, the minimum score is 35. For 4-point Likert scale answers: not at all possible (1 point), definitely possible (4 points); For 5-point Likert scale answers: strongly disagree (1 point), strongly agree (5 points). As the scale score increases, the RSO level increases. In the validity and reliability study of the scale, the Cronbach Alpha coefficient was found to be 0.89.
Stigma Scale for Mental Illnesses for Health Care Workers | For 2 weeks
  The scale, which was developed by Kassam et al. (2012) and whose Turkish validity and reliability study was conducted by Azazi (2021), consists of 20 items. It is a scale using a 5-point Likert type rating. These are: strongly disagree (1 point), disagree (2 points), neither agree nor disagree (3 points), agree (4 points), and strongly agree (5 points). The maximum score that can be obtained from the scale is 100 (most stigmatizing), the minimum score is 20 (least stigmatizing). As the scale score increases, the level of stigmatization increases. In the validity and reliability study of the scale, the Cronbach Alpha coefficient was found to be 0.79.

IPD SHARING:
Plan to Share IPD: No